CLINICAL TRIAL: NCT04685551
Title: Improving Survivorship Outcomes for African American and Latinx Cancer Survivors and Caregiver Dyads Through A Culturally Based Training Program for Underserved Health Professional Students
Brief Title: Improving Survivorship Among Minority Cancer Dyads
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CancerDyads
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cancer; Breast Cancer; Colon Cancer; Caregiver Burnout; Lung Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colonic Neoplasms; Caregiver Burden; Lung Neoplasms | interventions — Health Resources

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivorship Management among African American and Latinx Cancer Dyads (Experimental): This arm will implement a "one group pre-test and posttest" design to improve health outcomes of African American and Latinx cancer survivors and caregivers in collaboration with health professional students trained as Cancer Survivorship and Caregiver Leaders Aimed for Minority Populations (CSC LAMPs).
  Interventions: Behavioral: Change in knowledge, motivation, skills, and resources

INTERVENTIONS:
Behavioral: Change in knowledge, motivation, skills, and resources — Provide/enhance knowledge, modify attitudes, motivate and provide skills and resources to improve survivorship outcomes.

SUMMARY:
This proposed intervention centers on improving survivorship outcomes among African American and Latinx cancer survivor and caregiver dyads. As a result, there will be four major outcomes. First, as a result of partnership with minority social institutions (e.g. faith leaders), we will develop an in-depth culturally sensitive curriculum and survivorship care plan for Cancer Survivorship and Caregiver Leaders Aimed for Minority Populations (CSC LAMPs). Second, we will increase knowledge and skills by evaluating a comprehensive cancer survivorship training program designed for underserved health professional students. Third, the implementation of this program will improve survivorship outcomes among African American and Latinx cancer survivors with advanced stage cancer and their caregivers. Lastly, this study will build sustainability for underserved minorities with the training of 30 future healthcare providers as a valuable community resource for improving cancer survivorship outcomes. The long-term outcomes of the CSC LAMPs program will generate workforce capacity and diversity in cancer-based clinical practice, research, and community advocacy for underserved minority cancer survivors and caregivers.

ELIGIBILITY:
Aim 1 Focus Group for Cancer Survivors and Caregivers:

Inclusion Criteria

* Individuals ages 18 and older
* identify as African American or Latinx
* identify as a cancer survivor and/or caregiver
* speak and/or understand English

Exclusion Criteria

* individuals ages 17 years or younger
* does not identify as African American or Latinx
* unable to speak or understand English
* does not identify as a cancer survivor or caregiver

Aim 1 Focus Group for Oncology Healthcare Providers:

Inclusion Criteria

* Individuals ages 18 and older
* identify as a healthcare provider
* provide care to cancer patients in current provider role
* speak and/or understand English

Exclusion Criteria

* individuals ages 17 years or younger
* unable to speak or understand English
* does not provide care to cancer patients
* does not identify as a healthcare provider

Aim 2:

Inclusion Criteria

* Individuals ages 18 and older
* registered as a CDU student
* speak and/or understand English
* considered to be underserved, which include a) identifying as an underrepresented minority: Asian, Pacific Islander, African American, Hispanic, and Native American/Alaskan Native and/or b) from a medically underserved population (i.e. faced economic, cultural or linguistic barriers to health care)

Exclusion Criteria

* individuals ages 17 years or younger
* not registered as a CDU student
* unable to speak or understand English
* not considered to be underserved

For Aim 3:

Inclusion Criteria

* cancer survivor with a participating caregiver
* stage III or stage IV cancer diagnosis
* breast, lung, or colorectal cancer diagnosis
* identify as African American or Latinx
* speak and/or understand English

Exclusion Criteria

* individuals ages 17 years or younger
* does not identify as African American or Latinx
* unable to speak or understand English
* does not identify as a cancer survivor
* cancer survivor does not identify a caregiver
* does not have a breast, lung, or colorectal cancer diagnosis
* not diagnosed with a stage III or stage IV cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase in psychosocial well-being using the Quality of Life: Short Form Health Survey and the Center for Epidemiologic Studies Depression Scale | 3 months
  By comparison from baseline to post-intervention, there will be a 25% increase in the psychosocial well-being among study participants.
Reduction of barriers to symptom management Using the Symptom Distress Scale survey | 3 months
  By comparison from baseline to post-intervention, there will be a 25% decrease in the barriers to symptom management among study participants.
3. Decrease in unmet needs Using the Barriers to Follow-Up Care Survey and Cancer Survivors Unmet Needs instrument | 3 months
  By comparison from baseline to post-intervention, there will be a 25% decrease in the unmet needs among study participants.
Reduction in caregiver burden using the Caregiver reaction assessment (CRA) survey | 3 months
  By comparison from baseline to post-intervention, there will be a 25% decrease in the caregiver burden among study participants.
5. Increase knowledge and utilization of supportive services using the Medical Outcomes Study Social Support Survey | 3 months
  By comparison from baseline to post-intervention, there will be a 25% increase in the knowledge and utilization of supportive services among study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cobb, Principal Investigator — Charles R. Drew University of Medicine & Science
Locations (1):
- Charles R. Drew University of Medicine & Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No